CLINICAL TRIAL: NCT07014644
Title: A Randomized, Double-blind, Single-center Clinical Study to Evaluate the Efficacy and Safetyof Naltrexone Implant in Antagonizing Opioid Agonist Hydromorphone
Brief Title: A Randomized, Double-Blind, Single-Center Clinical Study on the Efficacy of Naltrexone Implant in Antagonizing Opioid Agonist Hydromorphone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen Sciencare Medical Industries Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HZ-Ⅱ-NQT-18-01
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.9 g (Experimental)
  Interventions: Drug: 0.9g Naltrexone Implant + 0.6g Naltrexone Implant Placebo
- 1.5 g (Experimental)
  Interventions: Drug: 1.5g Naltrexone Implant

INTERVENTIONS:
Drug: 0.9g Naltrexone Implant + 0.6g Naltrexone Implant Placebo — 0.9g Naltrexone Implant + 0.6g Naltrexone Implant Placebo
  Arms: 0.9 g
Drug: 1.5g Naltrexone Implant — 1.5g Naltrexone Implant
  Arms: 1.5 g

SUMMARY:
This study adopted a randomized, double-blind study design to evaluate the antagonistic effect, safety and pharmacokinetics of Naltrexone (opioid receptor antagonist) implantation after Hydromorphone (opioid receptor agonist) challenge.By using the method of multiple Hydromorphone challenge tests and assessing the clinical symptoms and signs related to opioid agonism as well as the pharmacokinetic parameters of Naltrexone and Hydromorphone, this study aimed to investigate the antagonistic effect of different doses of Naltrexone Implants post dosing in different time periods on different doses of Hydromorphone, to understand the ability of Naltrexone to antagonize Hydromorphone and its effective blood concentration, and to explore the effective dose and duration of Naltrexone Implants in antagonizing Hydromorphone. The study also aimed to provide a basis for the clinical use of Naltrexone Implants in the anti-relapse treatment of opioid dependence, and to provide a reference for the design of Phase 3 clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 65 years;
2. Those who had abused opioids for more than 1 year, and had used drugs at least once aweek in the abuse history;
3. Opioid-dependent subjects in the convalescent stage who had discontinued using opioids for more than 30 days and had a negative urine test for opioids;
4. Weight: male ≥ 45 kg, female ≥ 40 kg;
5. Physical condition: the subjects were screened within 2 weeks before the study, and had no medical history of heart, liver, kidney, digestive tract, nervous system, mental abnormality or metabolic abnormality; comprehensive physical examinations showed that the subjects had normal or abnormal but not clinically significant electrocardiogram, blood pressure, heart rate, respiratory status and laboratory tests including chest X-ray (results within half a year were valid), blood routine, urine routine, hepatic function, renal function, blood glucose, blood lipid, coagulation function and other biochemical tests at the discretion of the clinician;
6. Subjects without eye disease or optic neuropathy;
7. The subjects and their witnesses must give informed consent to this study before the study, and the subjects voluntarily signed a written informed consent;
8. The subjects could communicate well with the investigator and complete the study in accordance with the study regulations.

Exclusion Criteria:

* (1) Patients with clinically significant major diseases or major surgical operations within 4 weeks before the study; (2) Those with a history of heart, kidney, digestive tract and other important organs and hematopoietic system diseases; (3) Patients with bleeding tendency and leukopenia; (4) Patients with chronic pain or epilepsy; (5) Patients with serious mental and neurological diseases; (6) Patients with suicidal tendency; (7) Those who had a history of allergy to Hydromorphone or those who were allergic to Naltrexone and its excipients; (8) Those with blood loss or blood donation up to 200 ml within 3 months before the study; (9) Those who had participated in clinical studies of other drugs within 3 months before the study, or were participating in clinical studies of other drugs; (10) Those who had used drugs known to damage a certain organ or were currently using such drugs within 3 months before the study; (11) Those who had used prescription analgesics or psychiatric drugs within 30 days before the study; (12) Those who had used any drug that would inhibit or induce hepatic metabolism of drugs within one week before the study (e.g.: inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors - SSRI antidepressants, cimetidine, diltiazem macrolides, nitroimidazoles, sedative-hypnotics, verapamil, fluoroquinolones, antihistamines); (13) Any other surgical or medical condition that could potentially jeopardize the subject's participation in the study and alter the absorption, distribution, metabolism, and excretion of the drug, including the following:

  1. Inflammatory bowel syndrome, peptic ulcer, or gastrointestinal bleeding;
  2. History of serious gastrointestinal surgery, such as gastrectomy, gastrostomy, or colectomy;
  3. History of liver disease and hepatic function laboratory tests such as: alanine aminotransferase (ALT), aspartate aminotransferase (AST), γ-glutamyl transferase(γ-GT), or total bilirubin (T-Bili) greater than 1.5 × upper limit of normal (ULN) and judged by the clinician as abnormal and clinically significant；4) Clinically significant abnormalities in medical history or laboratory tests for creatinine, blood urea nitrogen, or urine components (e.g., proteinuria), suggesting renal impairment; (14) Those with a history of immunodeficiency, including a positive HIV test; (15) Those who were not suitable to participate in the study at the discretion of the investigator. In addition to the above requirements, female subjects who met the following conditions should also be excluded: (16) Those who took oral contraceptives 30 days before the study; (17) Those who had used within 6 months before the study and might use during the study long-acting estrogen or progestin injections or implants; (18) Women of childbearing age who had experienced unprotected sexual intercourse with their partners within 14 days before the study; (19) Women in pregnancy or lactating;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Effective Antagonistic Dose of Naltrexone Implant for Opioid Antagonism | 150 day
  Effective Antagonistic Dose of Naltrexone Implant for Opioid Antagonism

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University Address: No. 139, Renmin Road Central, Changsha City, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No